CLINICAL TRIAL: NCT01853267
Title: A Randomized Controlled Trial Evaluating the Requirement for Post-operative Packing of Perianal Abscesses
Brief Title: Perianal Abscess Packing Randomized ControlledTrial Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JRCOMS0513
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Perianal Abscess
Keywords: Colorectal; Surgery; Perianal; Abscess
MeSH Terms: conditions — Abscess | interventions — Control Groups; Drug Packaging

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Packing) (Active Comparator): The perianal abscess cavity will continue to be packed after discharge until healing is complete
  Interventions: Procedure: Control group (Packing)
- Intervention Group (Non-Packing) (Experimental): The cavity will be allowed to heal by secondary intention without packing.
  Interventions: Procedure: Intervention Group (Non-Packing)

INTERVENTIONS:
Procedure: Intervention Group (Non-Packing) — The haemostatic pack placed in the perianal abscess cavity will be removed on discharge and the wound will be left to heal without packing in situ
  Arms: Intervention Group (Non-Packing)
Procedure: Control group (Packing) — After the procedure the abscess cavity will be packed with a non-adherent dressing as per standard treatment and the packing changed at regular intervals in the community until healing by secondary intention is complete.
  Arms: Control group (Packing)

SUMMARY:
TITLE Perianal Abscess Packing (PAP): a randomised controlled trial (Pilot study)

DESIGN Randomised controlled trial.

HYPOTHESIS In patients with perianal abscesses incision and drainage without packing the subsequent cavity will reduce patient discomfort without increasing healing time or recurrence compared with management involving cavity packing.

OUTCOME MEASURES

* Length of hospital stay
* Time to cavity healing
* Recurrent abscess or fistula formation
* Pain score
* Analgesia usage POPULATION All patients older than 18 years presenting with a perianal abscess.

ELIGIBILITY Exclusion criteria:

* under 18 years
* those unable to give informed consent
* abscesses associated with Crohn's disease or other underlying causes
* abscesses in which initial drainage is considered inadequate (if the skin is not open sufficiently to allow drainage of the abscess cavity)

DURATION Until recruitment of subjects is complete

DETAILED DESCRIPTION:
1. INTRODUCTION

   1.1 BACKGROUND

   Perianal abscesses are common with an incidence of 0.5-1%. Some present as emergencies and all require surgery, placing a significant burden on health resources.

   The mainstay of management is incision and drainage. Traditionally the residual cavity is then packed. On discharge, the cavity packing requires frequent changing. This uses considerable community nursing resource. Perianal abscesses can alternatively be treated by primary closure or without packing the cavity. Benefits of treating without packing include greater patient comfort and acceptance and reduced nursing requirement. However treating without packing is not yet widely accepted, in the absence of sufficient evidence that it is as safe and effective. This study aims to address this issue.

   1.2 RATIONALE FOR CURRENT STUDY
   * Question: In patients with perianal abscesses, does incision and drainage without packing the subsequent cavity reduce patient discomfort without increasing healing time or recurrence compared with management involving cavity packing?
   * Hypothesis: Perianal abscess can be managed without cavity packing, with no increase in healing time or recurrence.
   * Note this was partly addressed by Tonkin et al (2004) but their study was underpowered. We intend to have a sufficiently powered study to definitively answer the question.
2. STUDY OBJECTIVES

   - Assess whether there is any statistically significant difference in patients with perianal abscesses managed with and without cavity packing in terms of:
   * Length of hospital stay
   * Time to cavity healing
   * Recurrent abscess or fistula formation
   * Pain score
   * Analgesia usage
3. STUDY DESIGN

   * This is a randomised controlled trial.
   * Due to the nature of the intervention (packing), it is impossible for either the subjects or the research team to be blinded.
   * Duration: recruitment into the study will remain open until the target number of subjects has been reached.
   * Number and type of subjects: power calculations from a published pilot study show that to demonstrate a difference of 10% vs 20% in e.g. fistula and recurrent abscess formation, 316 patients need to be recruited. We will perform a pilot study of 20 patients in each group and at this time calculate the number of subjects to be recruited

   3.1 STUDY OUTCOME MEASURES
   * Length of hospital stay
   * Time to cavity healing
   * Recurrent abscess or fistula formation
   * Pain score
   * Analgesia usage
4. PARTICIPANT ENTRY

   4.1 PRE-REGISTRATION EVALUATIONS
   * Documentation of the duration of symptoms before presentation.
   * Examination and documentation of abscess characteristics (can be done at the time of the operation): size, site and type.
   * Comorbidities

   4.2 INCLUSION CRITERIA
   * Perianal abscess.
   * Over 18 years of age.

   4.3 EXCLUSION CRITERIA
   * Under 18 years of age.
   * Those unable to give informed consent.
   * Abscesses associated with Crohn's disease or other underlying causes.
   * Abscesses in which initial drainage is considered inadequate (if the skin is not open sufficiently to allow drainage of the abscess cavity).

   4.4 WITHDRAWAL CRITERIA
   * If the patient wants to withdraw from the study at any point they can do so and resume standardized treatment pathways
5. ADVERSE EVENTS

   5.1 DEFINITIONS Adverse Event (AE): any untoward medical occurrence in a patient or clinical study subject.

   Serious Adverse Event (SAE): any untoward and unexpected medical occurrence or effect that:

   • Results in death
   * Is life-threatening - refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe
   * Requires hospitalization, or prolongation of existing inpatients' hospitalization
   * Results in persistent or significant disability or incapacity
   * Is a congenital anomaly or birth defect

   Medical judgement should be exercised in deciding whether an AE is serious in other situations. Important AEs that are not immediately life-threatening or do not result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes listed in the definition above, should also be considered serious.

   5.3 REPORTING PROCEDURES All adverse events should be reported. Depending on the nature of the event the reporting procedures below should be followed. Any questions concerning adverse event reporting should be directed to the Chief Investigator in the first instance.
6. ASSESSMENT AND FOLLOW-UP

   - Patients in the packing group will have their dressing changed day 1 post-operatively. On discharge they will have their care transferred to the District Nurses for daily dressing care in their own home.
   * Patients in the non-packing group will have the initial haemostatic dressing removed day 1 post-operatively and be discharged with a superficial protective dressing to absorb any discharge and protect the wound.
   * All patients will be reviewed at 2 weekly intervals in the outpatient clinic until the cavity is closed and the skin completely re-epithelialized. At outpatient appointments, patients will be asked to score their pain over the previous two weeks on a standard 10cm Visual Analogue Scale for pain.
   * Patients who do not attend clinic will be interviewed by telephone to gather the information listed above.
   * The end point is patient discharge from the outpatient clinic with complete healing (as described above) or the development of a fistula or recurrent abscess.
7. STATISTICS AND DATA ANALYSIS

   * Data and all appropriate documentation will be stored for a minimum of 5 years after the completion of the study, including the follow-up period.
   * The data will be tested for normal distribution and analyzed accordingly:

     o If it is normally distributed, an unpaired T-test will be performed on the continuous data (time to healing, length of stay, pain score, morphine dose) and a Fischer test will be performed on the categorical data (fistula rates, recurrence, delayed healing).
     * If it is not normally distributed, a Mann-Whitney U test will be performed in place of the T-test.
     * The tests will be two-tailed with a significance level of 0.05.
   * Following a pilot study of 40 patients we will perform a power calculation however a similar pilot study already published indicates the need for 316 subjects to be recruited

8.1 CONSENT Consent to enter the study must be sought from each participant only after a full explanation has been given, an information leaflet offered and time allowed for consideration. Signed participant consent should be obtained. The right of the participant to refuse to participate without giving reasons must be respected. After the participant has entered the study the clinician remains free to give alternative treatment to that specified in the protocol at any stage if he/she feels it is in the participant's best interest, but the reasons for doing so should be recorded. In these cases the participants remain within the study for the purposes of follow-up and data analysis. All participants are free to withdraw at any time from the protocol treatment without giving reasons and without prejudicing further treatment.

8.2 CONFIDENTIALITY The Chief Investigator will preserve the confidentiality of participants taking part in the study and is registered under the Data Protection Act.

8.3 AUDITS The study may be subject to inspection and audit by Imperial College London under their remit as sponsor and other regulatory bodies to ensure adherence to GCP and the NHS Research Governance Framework for Health and Social Care (2nd edition).

9. STUDY MANAGEMENT

The day-to-day management of the study will be coordinated through Mr Mikael Sodergren.

10. PUBLICATION POLICY

All publications and presentations relating to the study will be authorized by the Trial Management Group (TMG). The first publication of the trial results will be in the name of the Trial Management Group, or appropriately names authors. If there are named authors, these will include at least the trial's Chief Investigator, and Trial Coordinator. Members of the TMG will be listed and contributors will be cited by name if published in a Joint Research Office journal where this does not conflict with the journal's policy. Authorship of parallel studies initiated outside of the Trial Management Group will be according to the individuals involved in the project but must acknowledge the contribution of the Trial Management Group and the Study Coordination Centre.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18
* Clinical diagnosis of perianal abscess.

Exclusion Criteria:

* Patients who are unable or unwilling to consent.
* Known fistulae
* Crohn's Disease
* Immune-suppression or malignancy
* Recurrent abscess (where initial drainage insufficient).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Time to abscess healing | Two weeks post operative
  When abscess cavity has re-epitheliased. Assessed at two weeks and then weekly until healing occurs. Followed up for one year to assess recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Paraskevas Paraskevas, MBBS, Principal Investigator — Department of Surgery and Cancer, Imperial College London
Locations (1):
- St Mary's Hospital, Paddington, London, United Kingdom

REFERENCES:
- [Derived] Perera AP, Howell AM, Sodergren MH, Farne H, Darzi A, Purkayastha S, Paraskeva P. A pilot randomised controlled trial evaluating postoperative packing of the perianal abscess. Langenbecks Arch Surg. 2015 Feb;400(2):267-71. doi: 10.1007/s00423-014-1231-5. Epub 2014 Jul 23. PMID 25053508